CLINICAL TRIAL: NCT02198755
Title: Sensitivity, Specificity and Predictive Value of High Resolution (B-Mode) Ultrasonography (HRUS) for the Detection of Osteomyelitis in Chronic Wound Patients
Brief Title: Detection of Osteomyelitis Using High Resolution Ultrasound
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Calvary Hospital, Bronx, NY (Other)
Responsible Party: Principal Investigator, Oscar M. Alvarez, PhD, Director, Center for Curative and Palliative Wound Care, Calvary Hospital, Bronx, NY
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 100-Osteo-HRUS-0601
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Osteomyelitis
Keywords: high resolution ultrasound; osteomyelitis
MeSH Terms: conditions — Osteomyelitis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High Resolution Ultrasound (Active Comparator): High Resolution Ultrasonography (HRUS) with a Hitachi-Aloka Noblus Scanner
  Interventions: Device: Hitachi-Aloka Noblus ultrasound scanner
- Magnetic Resonance Imaging (MRI) (Active Comparator): Magnetic Resonance Imaging (MRI)
  Interventions: Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Device: Hitachi-Aloka Noblus ultrasound scanner — High resolution ultrasound with the Hitachi-Aloka Noblus Scanner and a 8-15mHz transducer
  Arms: High Resolution Ultrasound
Device: Magnetic Resonance Imaging (MRI) — MRI with or without contrast
  Arms: Magnetic Resonance Imaging (MRI)

SUMMARY:
The purpose of this study is to establish the sensitivity of HRUS as compared to MRI for the diagnosis of osteomyelitis in chronic wound patients; and to determine the specificity of HRUS as compared to pathologic and microbiologic studies of bone biopsy tissues.

ELIGIBILITY:
Inclusion Criteria:

1. Patient may be of any race and between 18-85 years of age.
2. Patient has a current diagnosis of a chronic ulcer with suspected osteomyelitis.
3. Patient's ulcer may be due to any etiology including but not limited to diabetes, trauma, neuropathic, pressure, venous, arterial, and inflammatory.
4. Patient's ulcer may extend through the dermis and into subcutaneous tissue (granulation tissue may be present), and may include exposure of muscle, tendon, bone, or joint capsule.
5. Patient's ulcer is suspected of causing a bone infection.
6. Patient's ulcer may be of any size.
7. Patient's wound may present with non-viable tissue.
8. Patient circulation to the wound should be evaluated and treated using normal protocol.
9. Patient's diabetes is under control as determined by the Investigator. Patients must have an HbA1c value less than 13.0%. Those patients whose glucose level is not deemed to be in control should be referred to their primary physician for treatment of the hyperglycemia.
10. Patient and caregiver are willing to participate in the clinical study and comply with the follow-up regimen.
11. Patient or his/her legal representative has read and signed the Institutional Review Board (IRB) approved Informed Consent form before treatment.
12. If patient is capable of childbirth, she is using medically accepted means of birth control, and she tests negative on a serum pregnancy test.
13. Active localized acute wound infection or cellulitis: Subject may be considered for study enrollment after the signs and symptoms of acute infection have resolved.

Exclusion Criteria:

1. Subject has a condition where an MRI is contraindicated

   * Metallic fragments, clips or devices in the brain, eye, spinal canal, etc.: (Plain radiography is sufficient for screening
   * Magnetically activated implanted devices:

   Cardiac pacemakers, insulin pumps, neuro¬stim¬u¬lators, cochlear implants, etc. may be de-programmed.
   * Non-graphite spinal cord tongs: Graphite tongs are compatible.
   * Thermodilution Swan-Ganz catheter: Local heating can result. If unenhanced MRI is likely to provide sufficient information, gadolinium should not be administered to these patients. If, after review of clinical indications, gadolinium enhancement is judged to be important for diagnosis, the lowest effective dose of contrast agent should be used.
2. In subjects where gadolinium enhancement MRI is planned then the following exclusion criteria apply:

   * Subject is allergic to contrast materials or cannot tolerate gadolinium
   * Subject is at risk of nephrogenic systemic fibrosis (NSF) or has severe renal failure (as determined by the investigator)
3. Patient must not be pregnant.
4. Patient has any condition(s) that seriously compromises the patient's ability to complete this study.
5. Patient with recent surgical debridement of the bone in and around the ulcer site.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-12; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Percent sensitivity and specificity of HRUS as compared to MRI and bone biopsy | at 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Oscar M Alvarez, PhD, Principal Investigator — Director, Wound Care Center, Calvary Hospital; Martin Wendelken, DPM, RN, Study Director — Staff Podiatrist, Wound Care Center, Calvary Hospital, Bronx, NY
Locations (1):
- Center for Curative and Palliative Wound Care, Calvary Hospital, The Bronx, New York, United States